CLINICAL TRIAL: NCT00667329
Title: Primary Treatment of Macroglobulinemic Lymphoma With 2CdA, Cyclophosphamide and Rituximab
Brief Title: Treatment of Macroglobulinemic Lymphoma With 2CdA, Cyclophosphamide and Rituximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM99-070; NCI-2020-00334 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma
Keywords: Waldenstrom's Macroglobulinemia; Lymphoma; 2CdA; Cladribine; Leustatin; Cyclophosphamide; Cytoxan; Neosar; Rituxan; Rituximab
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Cladribine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 2CdA + Cyclophosphamide + Rituximab (Experimental): 2CdA 1.5 mg/m^2 subcutaneous injection three times daily x 7 days. Cyclophosphamide 40 mg/m^2 PO twice daily x 7 days. Rituximab 375 mg/m^2 IV once weekly x 4 weeks.
  Interventions: Drug: 2CdA; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: 2CdA — 1.5 mg/m^2 subcutaneous injection three times daily x 7 days.
  Other Names: Leustatin; Cladribine
Drug: Cyclophosphamide — 40 mg/m^2 PO twice daily x 7 days.
  Other Names: Cytoxan; Neosar
Drug: Rituximab — 375 mg/m^2 IV once weekly x 4 weeks.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to see how well the drugs 2CdA, cyclophosphamide, and rituximab (rituxan) shrink a lymphoma called Waldenstrom's macroglobulinemia. After these drugs are given for 2 courses, a second goal is to see how long a remission lasts. A third goal is to see how often repeat remissions can be achieved when the lymphoma returns later and the same drugs are restarted.

This is an investigational study. The FDA has approved each of these drugs for the treatment of low-grade lymphoma. The combined use of these drugs for Waldenstrom's macroglobulinemia is investigational, although each drug has been effective by itself for this disease. About 50 patients will take part in this study. This study will take place only at UTMDACC (outpatient basis).

DETAILED DESCRIPTION:
Before the study starts, patients will have a complete exam. Blood and urine tests will be done. A bone marrow test, a chest x-ray and a CT scan of the abdomen will be done if not studied recently.

Blood tests will be repeated after 14, 21, and 42 days. Provided the disease has responded, another bone marrow sample will be taken to confirm remission. X-rays may be repeated for the same reason.

The patient or a family member will be taught to inject 2CdA under the skin three times a day for 7 days. The patient will also take cyclophosphamide by mouth twice each day. Rituxan will be given by vein once weekly for 4 weeks after a test infusion on the day prior to the first injection. A second course of the 3 drugs will be given about 6 weeks after the start of the first course. All patients with improving disease will then be followed without further treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with symptomatic macroglobulinemic lymphoma are eligible. Macroglobulinemic lymphoma includes patients with either biopsy proven small lymphocytic lymphoma or chronic lymphocytic leukemia and monoclonal IgM. Also included are symptomatic patients with clonal proliferation producing a pathologic monoclonal IgM that causes cryoglobulinemia, peripheral neuropathy or cold agglutinin hemolytic anemia.
2. Patients must have adequate liver function (bilirubin <2.5 mg%) and renal function (creatinine <2.0 mg%).

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1999-07-09 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Response Rate | two months
  Response defined as at least 50% reduction of monoclonal IgM synthesis for at least two months with more than 50% reduction of tumor infiltrates at all involved sites (bone marrow, lymph nodes, spleen etc.). Complete response defined as disappearance of abnormal protein by immunofixation, resolution of lymphadenopathy and splenomegaly, less than 20% lymphocytes in bone marrow and no evidence of monoclonal lymphocytes.

SECONDARY OUTCOMES:
After these drugs are given for 2 courses, a second goal is to see how long a remission lasts. | 10 Years
A third goal is to see how often repeat remissions can be achieved when the lymphoma returns later and the same drugs are restarted. | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Donna M. Weber, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org